CLINICAL TRIAL: NCT03264872
Title: Peer-enhanced Motivational Interviewing for Emerging Adults With Risky Substance Use
Brief Title: Peer MI for Substance-using Emerging Adults
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Douglas Smith, Associate Professor, School of Social Work, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB17393
Record Dates: First submitted 2017-08-23; First posted 2017-08-29 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Substance-Related Disorders
Keywords: Motivational Interviewing
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-Enhanced Motivational Interviewing (Experimental): Both dyad members, the target client and their peer support person, in this Peer-Enhanced Motivational Interviewing arm will receive separate one-hour Motivational Interviewing (MI) sessions with a trained counselor.
  Interventions: Behavioral: Peer-Enhanced Motivational Interviewing
- Waitlist Control (Other): Delayed Treatment.
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Behavioral: Peer-Enhanced Motivational Interviewing — Target clients in this Peer-Enhanced Motivational Interviewing arm will receive separate one-hour Motivational Interviewing (MI) sessions, in which the therapist reviews the target clients substance use behaviors in a non-confrontational manner, listens empathetically, and reinforces any client statements indicating a desire the change. In this arm, the therapist also presents the target client's peer with data about the extent of the target client's substance use, builds the peer's motivation to help their friend, and teaches the peer communication sills they can use to influence the target client's substance use behaviors.
  Arms: Peer-Enhanced Motivational Interviewing
Other: Waitlist Control — After the 12 week follow up period, if subjects in the Waitlist Control group desire to receive the Peer-Enhanced Motivational Interviewing intervention, that will be made available to them.
  Arms: Waitlist Control

SUMMARY:
The main purpose of this project is to test whether Peer-Enhanced Motivational Interviewing (PMI) results in superior alcohol and marijuana use outcomes for emerging adults (EAs, ages 18-29) and their peers. Ninety peer dyads (total n = 180, ntarget client = 90, npeer = 90) are randomized to receive either Peer-Enhanced Motivational Interviewing (PMI) or Waitlist Control (WC).

DETAILED DESCRIPTION:
This project randomized peer dyads, consisting of one EA (Emerging Adult; 18-29 years old) with a substance use problem (i.e. target client) and one peer, to one of two conditions. In the Peer-Enhanced Motivational Interviewing (PMI) condition, target clients and peers will receive separate one-hour sessions of Motivational Interviewing (MI) , an empirically-supported treatment that helps individuals work through ambivalence about making changes in substance use. MI is thought to work because it is a non-confrontational intervention where a therapist empathetically reviews substance use behaviors, listens empathetically, and reinforces any client statements indicating a desire to change. With the 'peer' of each PMI dyad, the therapist presents peers with data about the extent of the target client's substance use, builds the peer's motivation to help their friend, and teaches the peer communication skills they can use to influence the target client's substance use. In the WC condition, target clients and peers can receive PMI after the study follow-up period. Both target clients and their peers are followed for 12 weeks post-intervention.

The main purpose of this project is to test whether Peer-Enhanced Motivational Interviewing (PMI) results in superior alcohol and marijuana use outcomes for emerging adults (EAs, ages 18-29) and their peers. Ninety peer dyads (total n = 180, ntarget client = 90, npeer = 90) are randomized to receive either Peer-Enhanced Motivational Intervie (PMI) or Waitlist Control (WC).

ELIGIBILITY:
Inclusion Criteria:

For the Target Client

* Score 5 or higher on the AUDIT-C measure and/or use alcohol or marijuana 13 days or more out of the past 90 days,
* Have a friend that they are willing to refer to the study to be their 'peer' (support) and that peer agrees to participate,
* Are able to complete baseline and follow-up assessments and have a valid email,
* Are willing to be video recorded, and
* Are fluent in English

For the Peer

* Have weekly contact with the participating Target Client who referred them,
* Are will to attend all study procedures (i.e. baseline assessment, intervention, follow up),
* Are willing to be video record,
* Are fluent in English

Exclusion Criteria:

For the Target Client

* Are current students in the lead Investigator's classes,
* Are seeking residential treatment at the time of the screening call,
* Are incarcerated or court-ordered to receive treatment at the time of the screening call,
* Use drugs besides marijuana or alcohol over 45 of the past 90 days.

For the Peer

* Are current students in the lead Investigator's classes,
* Are seeking residential treatment at the time of the screening call,
* Are incarcerated or court-ordered to receive treatment at the time of the screening call,
* Use drugs besides marijuana or alcohol over 45 of the past 90 days,
* Are romantic partners of the Target Client

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-03-08 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
GAIN Substance Problem Scale | Baseline and every 2 weeks during 12 week post-intervention period
  a 16-item scale composed of lifetime symptoms of substance abuse, dependence, and substance-induced health and psychological disorders based on the DSM-IV

SECONDARY OUTCOMES:
GAIN Substance Frequency Scale (change) | Baseline and every 2 weeks during 12 week post-intervention period
  The GAIN substance frequency scale (SFS) measures the percent of days of substance use and percent of days of related problems from such substance use. This scale encompasses a large number of classes of substances, found to be ideal for measurement among poly- substance using individuals.
Rutgers Alcohol Problem Index (change) | Baseline and every 2 weeks during 12 week post-intervention period
  a 23-item self-administered screening tool (questionnaire) for assessing adolescent problem drinking. Respondents simply circle the number that corresponds to the number of times they have experienced each problem. Items can also be read aloud by an interviewer to clients with reading difficulties or it can be used as a springboard for a discussion of problems related to the client's alcohol use.
Significant Other Behavior Questionnaire | Baseline and every 2 weeks during 12 week post-intervention period
  An instrument measuring the specific social support in terms of the patient's drinking. Assessments of the significant other's behavior in the presence of the patient drinking is provided by both the patient and significant other.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas C Smith, PhD, Principal Investigator — University of Illinois Urbana Champaign School of Social Work
Locations (1):
- School of Social Work, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No